CLINICAL TRIAL: NCT03381534
Title: Safety and Efficacy of Distal Embolic Protection Device in Vertebral Artery Origin Stent Angioplasty :A Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Safety and Efficacy of Distal Embolic Protection Device in Vertebral Artery Origin Stenting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, lingfeng, director of neurosurgery department of Xuanwu hospital, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XuanwuH-VAO
Record Dates: First submitted 2017-05-26; First posted 2017-12-22 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Adverse Event
Keywords: vertebral artery origin; angioplasty; distal embolic protection
MeSH Terms: interventions — Stents

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stent assisted angioplasty (Placebo Comparator): patient randomly assigned to this group would be undergone stenting of vertebral artery origin without embolic protection device
  Interventions: Device: stent assisted angioplasty
- stenting with EPD (Experimental): patient randomly assigned to this group would be undergone stenting of vertebral artery origin with embolic protection device
  Interventions: Device: stenting with EPD

INTERVENTIONS:
Device: stenting with EPD — participants will be randomly assigned to control group or experimental group,patients in control group will be undergone stenting of vertebral artery origin without embolic protection device,patient in experimental group will be undergone stenting of vertebral artery origin with embolic protection device
  Arms: stenting with EPD
Device: stent assisted angioplasty — participants will be randomly assigned to control group or experimental group,patients in control group will be undergone stenting of vertebral artery origin without embolic protection device,patient in experimental group will be undergone stenting of vertebral artery origin with embolic protection device
  Arms: stent assisted angioplasty

SUMMARY:
This is a prospective single-center,randomized controlled trial,aiming to investigate the safety and efficacy of distal EPD in vertebral artery origin stenting(VAOS);256 subjects will be recruited in this study,after randomized recruitment, treatment group(128 subjects each group) undergo VAOS with adjuvant distal embolic protection device（EPD）,control group undergo routine VAOS without distal embolic protection device.Intraprocedural and postprocedural in-hospital adverse events,including stroke,death and dis-retrieval of EPD,will be noted and cost-effectiveness analysis also will be conduct,including economic cost,hospital stays.

DETAILED DESCRIPTION:
Ischemic cerebrovascular diseases are associated with a high rate of mortality and disability rate, as a consequence, many related trials were conducted to perfect prophylaxis and treatment of ischemic stroke. 2/3 of cerebral blood supply is offered by Internal carotid artery(ICA) , due to high morbility and disability rate of carotid territory stroke, stoke caused by ICA stenosis is always emphasized by authors. With the development to the depth in this field, ischemic stroke in posterior circulation related to vertebral artery stenosis is gradually paid attention recently. Outcome from New England medical center posterior circulation registry study revealed that 20% of patients were found to have vertebral artery origin(VAO) stenosis, in 9% of these patients, no other cause of stroke was identified. The relative risk of having a stroke or dying in patients with VAO stenosis was 6 times than that of patients without VAO stenosis. Therefore, VAO stenosis need appropriate management to prevent potentiality of ischemic stroke.

Nowadays there are three treatment alternatives for extracranial VAO stenosis: medicine, surgery and endovascular stent angioplasty. However, medical therapy mainly focus on prevention and delay of severe ischemic events other than radical therapy, and it's not always effective to improve symptoms of posterior circulation ischemia. Surgery are limited by its serious trauma and the combined postoperative morbidity and mortality rates ranging from 10% to 20%.Endovascular stent angioplasty was feasible in ICA stenosis as reported in literatures, and that promotes the utilization of stent in VAO stenosis in recent years. Related retrospective studies have demonstrated the safety and efficacy of vertebral artery origin stenting(VAOS) in VAO stenosis. In a Meta analysis that summarized 27 articles about extracranial vertebral artery stenting, Stayman observed that the rate of transient ischemic attack(TIA) and stroke within postprocedural 30 days was 1.1% and 0.8% respectively. Compter etc. are conducting a prospective case-control study to assess the safety and feasibility of VAOS, which final outcome is thought to be relatively authentic.

However, some drawbacks in VAOS needs additional resolution, like embolization caused by plaque debris, high restenosis rate, vasospasm, vessel dissection. Especially, embolization is associated with not only plaque characteristic, but also anatomy of the vertebral arteries, which is potentially essential to high risk of plaque debris dislodgment. The origin of vertebral artery is characterized with small diameter and tortuous course. Dodevski analyzed 30 patients' vertebral arteries and found that 40% of patients' vertebral artery was tortuous, the diameter of the VAO on the left side was in the range between 1.60-5.2 mm, mean 3.33 ± 0.89 mm, and on the right side from 1.64-5.40 mm, mean 3.19 ± 0.98 mm. Tortuosity and small diameter in VAO will increase operation difficulty and procedural time. Borhanisummarized 27 articles focusing on vertebral origin angioplasty and concluded that of the 808 patients underwent stent angioplasty, the combined rate of stroke and TIA within 1 month after stenting was 6.9%.

Concerning dislodgement of plaque debris, embolic protection device(EPD) is applied recently to decrease the risk of embolization. But utilization of EPD in VAOS is mainly based on its safety and feasibility in carotid artery stenting(CAS). In CAS, cerebral embolic protection devices can effectively reduce the incidence of transient ischemic attack, stroke and other related adverse events. The U.S. Safety Committee recommended stopping unprotected CAS, because the 30-day rate of stroke was 3.9 times higher than that of CAS with cerebral protection. However, VAOS is different from CAS, and its performance in CAS cann't serve as medical science evidence for distal EPD in VAOS. Firstly, the rate of postoperative restenosis after VAOS is higher than that of CAS, ranging from 20% to 66.7%.Secondly, VAO are characterized by concentric, fibrous, and smooth lesions with lower incidence of ulceration and intraluminal hemorrhage compared with extracranial carotid artery circulation[13]. Thirdly, the microscopic structure of VAO is featured with elastic fibers and smooth muscles. These distinctions indicate that investigators should make a distinction between CAS and VAOS in terms of intravascular intervention. As to the use of EPD in VAOS, no Class Ⅰ evidence can verify the safety and efficacy of EPD and clinicians share discrepant opinions. Some authors thought that distal protection devices will suspend operation process, increase operation-related risk and may cause embolization during crossing lesion and retrieval which may be referable to transient shear stress. In addition, some patients are intolerable to flow cessation caused by distal EPD. Moreover, foreign case reports even noted that utilization of distal EPD was probable to induce vasospasm and difficult retrieval of distal EPD was finally managed by secondary surgery in some cases[14, 15]. However, small sample-size studies demonstrated it's safe and feasible to use distal EPD in VAOS. Qureshi etc.retrospectively analyzed clinical data of 12 patients underwent VAOS with filter protection, outcome revealed that no stroke and death events occured within 1 month follow-up. In a multicenter study, Edgell etc. contrastively analyzed the data of patients underwent VAOS with and without distal EPD, the rate of TIA and stroke within 1 month between the two groups showed no significant difference. Divani etc. analyzed plaque debris captured by EPDs in 14 patients who underwent VAOS with distal protection devices, the outcome revealed that relative to the size of the filter, the proportion of captured debris ranged from 0.1% to 22% in the VA filters, hence, Divani recommended the use of distal EPD in VAOS.

In summary, the use of distal EPD in VAOS is debatable, no class I evidence can support the advantage of use of distal EPD in VAOS. Here, the investigators will conduct this prospective, single-center, randomize controlled trial aiming to analyzed the safety and efficacy of distal EPD in VAOS.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40 to 80 years old;
2. VAO atherosclerotic stenosis results in posterior circulation ischemic symptom refractory to best medical treatment;
3. symptomatic VAO atherosclerotic stenosis>70% evaluated by computed tomograph angiography(CTA) or Magnetic Resonance Angiography(MRA) or digital subtraction angiography(DSA);
4. the diameter of the normal segment of the artery beyond the stenosis >3.5mm;
5. written informed consent.

Exclusion Criteria:

1. VAO stenosis is combined with ipsilateral vertebrobasilar disease including severe cranial vertebral artery stenosis and severe basilar artery stenosis.
2. VAO is occluded;
3. Patients who will be underwent bilateral VAOS due to bilateral VAO stenosis including someone with bilateral VAO stenosis >70% and the patient who need contralateral VAOS after stenting in unilateral VAO due to recurrent posterior circulation ischemia refractory to best medical treatment.
4. VAO stenosis caused by arteritis,artery dissection, aplasia, vasculopathy caused by radiotherapy etc, other than atherosclerosis;
5. stroke within 30 days or myocardial infarction within 6 months;
6. contraindication of anticoagulant and antiplatelet agents; allergy to iodinated contrast agent;
7. severe comorbid diseases and intolerant to procedure; patient unlikely to cooperate with the procedure or provide informed consent.
8. High risk of difficulty or failure in EPD advance and retrieval due to the tortuosity of the culprit vertebral artery origin.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2017-05-20 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
embolus capture rate in patients treated with VAO stenting with EPD | during procedure
  embolus capture rate is calculate by number of patients with embolus in EPD divided number of patients without embolus in EPD in EPD group

SECONDARY OUTCOMES:
incidence of ischemic stroke in the two group | 30 days after procedure
  number of patients with or without ischemic stroke in posterior circulationcirculation territory will be collected in EPD group
incidence of disable or fatal ischemic stroke in EPD group | 1 month after procedure
  number of patients who present disable of fatal ischemic stroke in posterior

CONTACTS AND LOCATIONS:
Overall Officials: Jiao Li Qun, MD, Principal Investigator — Xuanwu Hospital of Capital Medical University
Locations (1):
- XuanWu hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wityk RJ, Chang HM, Rosengart A, Han WC, DeWitt LD, Pessin MS, Caplan LR. Proximal extracranial vertebral artery disease in the New England Medical Center Posterior Circulation Registry. Arch Neurol. 1998 Apr;55(4):470-8. doi: 10.1001/archneur.55.4.470. PMID 9561974
- [Result] Thompson MC, Issa MA, Lazzaro MA, Zaidat OO. The natural history of vertebral artery origin stenosis. J Stroke Cerebrovasc Dis. 2014 Jan;23(1):e1-4. doi: 10.1016/j.jstrokecerebrovasdis.2012.12.004. Epub 2013 Jan 16. PMID 23332862
- [Result] Stayman AN, Nogueira RG, Gupta R. A systematic review of stenting and angioplasty of symptomatic extracranial vertebral artery stenosis. Stroke. 2011 Aug;42(8):2212-6. doi: 10.1161/STROKEAHA.110.611459. Epub 2011 Jun 23. PMID 21700936
- [Result] Compter A, van der Worp HB, Schonewille WJ, Vos JA, Algra A, Lo TH, Mali WP, Moll FL, Kappelle LJ. VAST: Vertebral Artery Stenting Trial. Protocol for a randomised safety and feasibility trial. Trials. 2008 Nov 24;9:65. doi: 10.1186/1745-6215-9-65. PMID 19025615
- [Result] Edgell RC, Zaidat OO, Gupta R, Abou-Chebl A, Linfante I, Xavier A, Nogueira R, Alshekhlee A, Kalia J, Etezadi V, Aghaebrahim N, Jovin T. Multicenter study of safety in stenting for symptomatic vertebral artery origin stenosis: results from the Society of Vascular and Interventional Neurology Research Consortium. J Neuroimaging. 2013 Apr;23(2):170-4. doi: 10.1111/j.1552-6569.2011.00665.x. Epub 2011 Dec 30. PMID 22211776
- [Result] Hatano T, Tsukahara T, Miyakoshi A, Arai D, Yamaguchi S, Murakami M. Stent placement for atherosclerotic stenosis of the vertebral artery ostium: angiographic and clinical outcomes in 117 consecutive patients. Neurosurgery. 2011 Jan;68(1):108-16; discussion 116. doi: 10.1227/NEU.0b013e3181fc62aa. PMID 21099720
- [Result] Taylor RA, Siddiq F, Memon MZ, Qureshi AI, Vazquez G, Hayakawa M, Chaloupka JC. Vertebral artery ostial stent placement for atherosclerotic stenosis in 72 consecutive patients: clinical outcomes and follow-up results. Neuroradiology. 2009 Aug;51(8):531-9. doi: 10.1007/s00234-009-0531-x. Epub 2009 May 13. PMID 19437002
- [Result] Lin YH, Juang JM, Jeng JS, Yip PK, Kao HL. Symptomatic ostial vertebral artery stenosis treated with tubular coronary stents: clinical results and restenosis analysis. J Endovasc Ther. 2004 Dec;11(6):719-26. doi: 10.1583/04-1336.1. PMID 15615563
- [Result] Albuquerque FC, Fiorella D, Han P, Spetzler RF, McDougall CG. A reappraisal of angioplasty and stenting for the treatment of vertebral origin stenosis. Neurosurgery. 2003 Sep;53(3):607-14; discussion 614-6. doi: 10.1227/01.neu.0000079494.87390.28. PMID 12943577
- [Result] Dodevski A, Lazareska M, Tosovska-Lazarova D, Zhivadinovik J, Aliji V. Morphological characteristics of the first part of the vertebral artery. Prilozi. 2011;32(1):173-88. PMID 21822186
- [Result] Borhani Haghighi A, Edgell RC, Cruz-Flores S, Zaidat OO. Vertebral artery origin stenosis and its treatment. J Stroke Cerebrovasc Dis. 2011 Jul-Aug;20(4):369-76. doi: 10.1016/j.jstrokecerebrovasdis.2011.05.007. PMID 21729790
- [Result] Mas JL, Chatellier G, Beyssen B; EVA-3S Investigators. Carotid angioplasty and stenting with and without cerebral protection: clinical alert from the Endarterectomy Versus Angioplasty in Patients With Symptomatic Severe Carotid Stenosis (EVA-3S) trial. Stroke. 2004 Jan;35(1):e18-20. doi: 10.1161/01.STR.0000106913.33940.DD. Epub 2003 Dec 4. PMID 14657456
- [Result] Zavala-Alarcon E, Emmans L, Little R, Bant A. Percutaneous intervention for posterior fossa ischemia. A single center experience and review of the literature. Int J Cardiol. 2008 Jun 23;127(1):70-7. doi: 10.1016/j.ijcard.2007.05.006. Epub 2007 Jul 24. PMID 17651834
- [Result] Cardaioli P, Giordan M, Panfili M, Chioin R. Complication with an embolic protection device during carotid angioplasty. Catheter Cardiovasc Interv. 2004 Jun;62(2):234-6. doi: 10.1002/ccd.20061. PMID 15170718
- [Result] Bornak A, Milner R. Current debate on the role of embolic protection devices. Vasc Endovascular Surg. 2012 Aug;46(6):441-6. doi: 10.1177/1538574412452160. Epub 2012 Jun 21. PMID 22723261
- [Result] Qureshi AI, Kirmani JF, Harris-Lane P, Divani AA, Ahmed S, Ebrihimi A, Al Kawi A, Janjua N. Vertebral artery origin stent placement with distal protection: technical and clinical results. AJNR Am J Neuroradiol. 2006 May;27(5):1140-5. PMID 16687560
- [Result] Mintz EP, Gruberg L, Kouperberg E, Beyar R. Vertebral artery stenting using distal emboli protection and transcranial Doppler. Catheter Cardiovasc Interv. 2004 Jan;61(1):12-5. doi: 10.1002/ccd.10710. PMID 14696152
- [Result] Divani AA, Berezina TL, Zhou J, Pakdaman R, Suri MF, Qureshi AI. Microscopic and macroscopic evaluation of emboli captured during angioplasty and stent procedures in extracranial vertebral and internal carotid arteries. J Endovasc Ther. 2008 Jun;15(3):263-9. doi: 10.1583/07-2326.1. PMID 18540698
- [Result] Gensicke H, Zumbrunn T, Jongen LM, Nederkoorn PJ, Macdonald S, Gaines PA, Lyrer PA, Wetzel SG, van der Lugt A, Mali WP, Brown MM, van der Worp HB, Engelter ST, Bonati LH; ICSS-MRI Substudy Investigators. Characteristics of ischemic brain lesions after stenting or endarterectomy for symptomatic carotid artery stenosis: results from the international carotid stenting study-magnetic resonance imaging substudy. Stroke. 2013 Jan;44(1):80-6. doi: 10.1161/STROKEAHA.112.673152. Epub 2012 Dec 13. PMID 23238861